CLINICAL TRIAL: NCT03365804
Title: A New Spinal Brace Design Concept for the Treatment of Adolescent Idiopathic Scoliosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00054113
Record Dates: First submitted 2017-12-02; First posted 2017-12-07 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Ultrasound; Scoliosis; Orthoses; 3D Printing
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Printed Brace (Experimental): This group will receive 3D printed brace
  Interventions: Device: 3D Printed Brace
- Traditional Brace (No Intervention): This group will receive the traditional brace

INTERVENTIONS:
Device: 3D Printed Brace — All subjects' body shape will be scanned to generate sterolithography (STL) files for 3D printing.
  Arms: 3D Printed Brace

SUMMARY:
Adolescent Idiopathic Scoliosis (AIS) is a three-dimensional deformity of the spine due to an unknown cause. Bracing is a proven non-surgical treatment for scoliosis. Our group developed an ultrasound assisted method which can improve brace design. However, it is still quite time consuming to construct a brace. Although 3D printing technology has been proposed to construct a scoliosis brace, its effectiveness has not been validated. The goals of this study was to investigate if an effective and comfortable brace can be designed and fabricated by using ultrasound and computer-aided design and computer-aided manufacturing (CAD/CAM) technology, and be printed directly from a 3D printer with faster production, lower cost, and improved comfort to patients. Also, to investigate the effectiveness of new designed brace. The final outcomes may reduce the total number of spinal surgeries for scoliosis. The benefits not only reduce the health care cost, but also increase the quality of life of these adolescent patients.

DETAILED DESCRIPTION:
A randomized clinical trial with a total of 50 new brace candidates diagnosed with AIS from the Stollery Children's Hospital Scoliosis Clinic will be conducted in the next 2 years. Ethics approval (Pro00054113) has been granted. Inclusion is based on the standard Scoliosis Research Society (SRS) brace studies criteria: a) diagnosed with AIS and new to rigid spinal brace treatment, b) prescribed full-time brace wear (23 hours per day), c) primary Cobb angles 20°- 40°, d) age between 10 -16 years, e) Risser 0-2 (skeletally immature), f) either premenarchal or less than 1 year postmenarchal. The 50 subjects will be randomly assigned to 2 equally sized groups (n=25 in each group): group A conventional designed and manual fabricated braces and group B ultrasound and CAD/CAM scanner designed brace with printing by a 3D printer.

Both groups: A brace monitor (2.5cm x 4.0cm x 1.5 cm and 8g) developed from our group will be installed into all braces for both study groups. It will monitor patients' compliance which includes how much time they use their braces and how much time they wear their braces at the prescribed tightness level (quantity and quality). The battery power and memory capacities of the monitor last for 9 months with the sample rate at 1 sample/minute. The brace monitor will be embedded into the brace). No extra attention is needed from the patients. The brace wear pattern data will be downloaded at the routinely scheduled follow up clinics (post brace prescription of 2 months, 6 months, 1 year and every 6 months periods).

For the compliance assessment, we will get 80% power in this sample size if the average compliance from the control group is 60±4% (from our previous study), but in the intervention group the compliance is increased to 70±4%. The compliance is the number of brace wear hours relative to the prescribed hours per day wear time.

Outcomes: When subjects return to their regular follow up scoliosis clinics, the standard standing in-brace radiographs will be taken. The in-brace Cobb angle will be measured by the clinic staff and saved into the clinical database. The Cobb angle correction (in percent) of the treated curve as measured at the immediate follow-up clinic (in-brace radiographic clinic) [(Pre-Out of brace Cobb angle - In-brace Cobb angle)/Pre-brace Cobb angle]*100 will be used to evaluate the immediate effectiveness. An unpaired 2-tailed Student's t-test using an alpha of 0.05 will be used to compare the correction observed in the intervention group to that of the control group. The total numbers of in-brace radiographs will be tailed; it will be counted up to the last radiograph that shows an in-brace correction which is deemed acceptable by the attending orthopedic surgeon. The number of radiographs will be compared between the two study groups. The p-value of the chi-squared test for independence will be used to determine whether a statistically significant difference exists between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

It is based on the standard SRS brace studies criteria: a) diagnosed with AIS and new to rigid spinal brace treatment, b) prescribed full-time brace wear (23 hours per day), c) primary Cobb angles 20°- 40°, d) age between 10 -16 years, e) Risser 0-2 (skeletally immature), f) if female either premenarchal or less than 1 year postmenarchal.

Exclusion Criteria:

* no surgery

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the in-brace Cobb angle on radiograph | It will be completed 2 months after the last participant is recruited.
  The in-brace Cobb angle will be measured from the radiograph at the first follow-up clinic.

SECONDARY OUTCOMES:
Evaluate participants' compliance on how they use their braces | The result can be reported within 6 months after the last participant is recruited.
  The data inside the brace monitors will be downloaded at each clinic visit to understand how well the participants use their brace. The time and wear tightness are the 2 parameters to be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Edmond Lou, PhD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No